CLINICAL TRIAL: NCT02683265
Title: A Randomized, Double-Blind, Placebo-Controlled, Flexible-Dose Titration Study of Aptensio XR® in Children Ages 4 to Under 6 Years Diagnosed With Attention Deficit-Hyperactivity Disorder (ADHD)
Brief Title: A Flexible-Dose Titration Study of Aptensio XR in Children Ages 4 to Under 6 Years Diagnosed With ADHD
Acronym: EF003
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RP-BP-EF003
Record Dates: First submitted 2016-02-05; First posted 2016-02-17 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Flexible-Dose Titration Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded active capsules looked identical to the same strength placebo capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aptensio XR (Experimental): Optimized dose of Aptensio XR (10, 15, 20, 30 or 40 mg Aptensio XR)
  Interventions: Drug: Aptensio XR
- Placebo comparator (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aptensio XR — Optimized dose of Aptensio XR (10, 15, 20, 30 or 40 mg) administered orally, once daily
  Other Names: methylphenidate, extended release
  Arms: Aptensio XR
Drug: Placebo — Placebo capsules
  Other Names: Dose-matched placebo
  Arms: Placebo comparator

SUMMARY:
This randomized, double-blind, flexible-dose, placebo-controlled, parallel group study is designed to evaluate Aptensio XR® compared to placebo in preschool age children with ADHD. Male and female children ages 4 years, 0 months to 5 years, 8 months with a diagnosis of ADHD (combined, inattentive or hyperactive/impulsive) will be enrolled.

There will be 6 phases in this study: a screening phase of up to 4 weeks, which will include washout if applicable, an enrollment & parent training phase lasting 2-4 weeks, an eligibility phase of up to 2 weeks to determine eligibility for the open-label phase, a 6-week open-label dose titration phase, a 2 week double-blind phase for Aptensio XR® responders, and a two-week follow-up call after study completion or early discontinuation to assess for ongoing adverse events and concomitant medications.

Up to 150 subjects will be enrolled in this trial to allow for subjects who improve significantly during the behavior training phase and drop-outs. Once 74 subjects have completed the double-blind phase, no additional subjects will be enrolled in the trial. Subjects who are already enrolled at that time will be allowed to complete the trial.

The primary objective of this study is to establish that an optimal dose of Aptensio XR® will result in a significant reduction in ADHD symptoms compared with placebo in children ages 4 to under 6 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ages 48 months to 68 months inclusive at time of consent
2. Met Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for ADHD, combined, hyperactive/impulsive or inattentive presentation made during a clinical interview by an experienced clinician and confirmed with Kiddie-Sads-Present and Lifetime Version (K-SADS-PL)
3. ADHD symptoms must have been present for at least 6 months
4. Age- and sex-adjusted ratings of ≥ 90th percentile Total Score on the ADHD-RS-IV Preschool Version
5. Score of < 65 on the Child Global Assessment Scale (CGAS)
6. Must have had a CGI-S score of ≥ 4 at Visit 2 (subjects who were granted a waiver to bypass parental training, and did not have a Visit 2, were still qualified to continue in the study based on their CGI-S score at screening)
7. Estimated intelligence quotient (IQ) ≥ 80 on the Kaufman Brief Intelligence Test, 2nd edition (KBIT-2). If results from the KBIT-2 were deemed invalid because of significant ADHD symptomatology, the PI could submit additional documentation to support average cognitive functioning. This documentation could include progress reports from preschool or other previous testing. These exceptions were evaluated by the Medical Monitor and Study PIs on a case-by-case basis for inclusion.
8. The subject had a parent or legal guardian who would give written informed consent for the subject to participate in the study
9. Subject and parent or legal guardian must have been able to speak and understand English
10. Subject must live with primary caretaker/rater and have been living with primary caretaker for at least 6 months
11. Subject and parent/guardian must have been willing and able to comply with all requirements of the protocol
12. Systolic and diastolic blood pressure below the 95th percentile for age and gender

Exclusion Criteria:

1. The subject had a lack of response to a trial of adequate dose and duration of MPH or intolerance to previous methylphenidate (MPH) treatment
2. The subject was using any other current psychotropic medication except clonidine, guanfacine, atomoxetine and/or stimulants or had taken an investigational drug in the 30 days prior to screening
3. The subject had used monoamine oxidase inhibitors (MAOIs) within 14 days of the screening visit
4. The subject planned to use prohibited drugs or agents at any point between the screening visit and the end of the study
5. Use of anticonvulsants, antidepressants, or antipsychotics in the 30 days prior to screening
6. The subject should not plan to start any additional psychotherapy outside of the trial during the duration of the study
7. The subject had a history of chronic vocal or motor tics or Tourette's syndrome
8. The subject had any clinically significant ECG abnormalities at screening
9. The subject had any major medical conditions that would have interfered with involvement in the study or could have been affected negatively by methylphenidate
10. The subject had chronic medical illnesses including a seizure disorder (excluding a history of febrile seizures), severe hypertension, untreated thyroid disease, known structural cardiac abnormalities, serious arrhythmias, cardiomyopathy, glaucoma, or a family history of sudden death
11. History (in the past 12 months) or presence of clinically-significant cardiovascular, cerebrovascular, renal, hepatic, gastrointestinal, pulmonary, immunological, hematological, endocrine, or neurological disease that in the opinion of the investigator could have put the subject at risk if he/she participated in the trial or which could have confounded study results
12. Family history (parent or sibling) of structural cardiovascular disease
13. Current or recent (past 12 months) history of drug abuse in someone living in the subject's home
14. Current symptoms or history of major psychiatric illness (for example schizophrenia, psychosis, bipolar disorder, post-traumatic stress disorder, depression, severe anxiety disorder, obsessive compulsive disorder or autistic spectrum disorder) in addition to ADHD that required treatment with additional medication or, in the opinion of the PI, would have contraindicated study participation
15. History or presence of suicidal ideation or significant self-injurious behavior
16. The subject showed evidence of current physical, sexual, or emotional abuse
17. Both biological parents of the subject had a history of bipolar disorder

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, MD, Principal Investigator — Center for Psychiatry And Behavioral Medicine Inc.
Locations (2):
- United States (2):
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7047252/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Enrolled Population consisted of all subjects who were not screen failures. Of these enrolled subjects, 119 entered the Open-label Treatment Phase and 90 were randomized to the Double-blind Treatment Phase.
Groups:
- Open-label Treatment Phase: 6-week open-label treatment phase. Aptensio XR capsules administered orally, once daily.
- Aptensio XR: Optimized dose of Aptensio XR administered orally, once daily.
- Placebo Comparator: Placebo capsules administered orally, once daily.
Period: Open-label Treatment Phase
Arm/Group | Open-label Treatment Phase | Aptensio XR | Placebo Comparator
Started | 119 | 0 | 0
Completed (The number who completed the Open-label Treatment Phase were randomized to 1 of 2 groups in the Double-blind Treatment Phase.) | 90 | 0 | 0
Not Completed | 29 | 0 | 0
Period: Double-blind Treatment Phase
Arm/Group | Open-label Treatment Phase | Aptensio XR | Placebo Comparator
Started | 0 | 40 | 50
Completed | 0 | 38 | 48
Not Completed | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aptensio XR | Placebo Comparator | Total
Number analyzed (Participants) | 40 | 50 | 90
Age, Continuous [Mean (Standard Deviation); unit: months] | 58.5 (5.59) | 59.2 (6.42) | 58.9 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 39 | 68
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 18 | 33
  White | 24 | 30 | 54
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Attention Deficit Hyperactivity Disorder Rating Scale - 4th Edition (ADHD-RS-IV) Preschool Version Total Score Change From End of Open Label Phase (Baseline) to End of Double Blind.
Description: ADHD-RS-IV is 18-item scale incorporates each of the ADHD symptoms listed in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) regardless of assigned subtype. Scoring was based on the universally accepted symptom severity as recommended in the DSM-IV-TR manual on a 4-point scale: 0 = never or rarely, 1 = sometimes, 2 = often, and 3 = very often. The total score is the sum of the scores for all 18 items and could range from 0 (no impairment) to 54 (maximal impairment) for each administration per subject. Higher score means higher frequency and severity of symptoms.
  Trained clinicians administered the questionnaire to parents. The ADHD-RS-IV Preschool Version was used to determine eligibility, optimal dosing and the efficacy of double blind treatment.
Time Frame: 2 weeks: End of open label phase (Baseline) at study day 84 to end of double blind treatment at study day 98.
Population: The Efficacy Evaluable (ITT-E) population consists of all subjects in the intent-to-treat (ITT) population who completed ADHD-RS-IV assessments at the end of the open-label treatment phase (i.e., baseline) and had at least one post-baseline ADHD-RS-IV assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aptensio XR | Placebo Comparator
Number analyzed (Participants) | 39 | 49
score on a scale | 6.3 (12.26) | 17.3 (16.76)

2. Secondary Outcome: Attention Deficit Hyperactivity Disorder Rating Scale - 4th Edition (ADHD-RS-IV) Preschool Version Hyperactivity-Impulsivity Subscale Score Change From End of Open Label Phase (Baseline) to End of Double Blind.
Description: This 18-item scale incorporates each of the ADHD symptoms listed in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) regardless of assigned subtype. Scoring was based on the universally accepted symptom severity as recommended in the DSM-IV-TR manual on a 4-point scale: 0=never or rarely, 1=sometimes, 2=often, and 3=very often. The Hyperactivity-Impulsivity even items. The Hyperactivity-Impulsivity subscale score was the sum of the scores for the 9 even items and could range from 0 (no impairment) to 27 (maximal impairment) for each administration per subject. Higher score means higher frequency and severity of symptoms.
  Trained clinicians administered the questionnaire to parents.
Time Frame: 2 weeks: End of open label phase (Baseline) at study day 84 to end of double blind treatment at study day 98.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aptensio XR | Placebo Comparator
Number analyzed (Participants) | 39 | 50
score on a scale | 3.36 (6.434) | 9.37 (8.762)

3. Secondary Outcome: Attention Deficit Hyperactivity Disorder Rating Scale - 4th Edition (ADHD-RS-IV) Preschool Version Inattention Subscale Score Change From End of Open Label Phase (Baseline) to End of Double Blind.
Description: This 18-item scale incorporates each of the ADHD symptoms listed in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) regardless of assigned subtype. Scoring was based on the universally accepted symptom severity as recommended in the DSM-IV-TR manual on a 4-point scale: 0=never or rarely, 1=sometimes, 2=often, and 3=very often. The Inattention subscales were based upon the sum of the odd items. The Inattention subscale score was the sum of the scores for the 9 odd items and could range from 0 (no impairment) to 27 (maximal impairment) for each administration per subject. Higher score means higher frequency and severity of symptoms.
  Trained clinicians administered the questionnaire to parents.
Time Frame: 2 weeks: End of open label phase (Baseline) at study day 84 to end of double blind treatment at study day 98.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aptensio XR | Placebo Comparator
Number analyzed (Participants) | 39 | 49
score on a scale | 2.9 (6.48) | 7.9 (8.48)

4. Secondary Outcome: Summary of Clinical Global Impression Scale of Severity (CGI-S) Score From End of Open Label Phase (Baseline) to End of Double Blind.
Description: The scale provides a global rating of illness severity during the trial. The subject is rated relative to the clinician's past experience with other subjects who have the same diagnosis. The CGI-S scale is 1 question and rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill subjects). A lower value a better the outcome.
Time Frame: 2 weeks: End of open label phase (Baseline) at study day 84 to end of double blind treatment at study day 98.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aptensio XR | Placebo Comparator
Number analyzed (Participants) | 39 | 50
Participants
  Baseline: 1 = Normal, not at all ill | 7 | 13
  Baseline: 2 = Borderline mentally ill | 15 | 14
  Baseline: 3 = Mildly ill | 8 | 11
  Baseline: 4 = Moderately ill | 7 | 11
  Baseline: 5 = Markedly ill | 1 | 1
  Baseline: 6 = Severely ill | 1 | 0
  Baseline: 7 = Among the most extremely ill subjects | 0 | 0
  End of Double-blind Treatment: 1 = Normal, not at all ill | 4 | 3
  End of Double-blind Treatment: 2 = Borderline mentally ill | 12 | 5
  End of Double-blind Treatment: 3 = Mildly ill | 5 | 4
  End of Double-blind Treatment: 4 = Moderately ill | 6 | 10
  End of Double-blind Treatment: 5 = Markedly ill | 10 | 19
  End of Double-blind Treatment: 6 = Severely ill | 2 | 7
  End of Double-blind Treatment: 7 = Among the most extremely ill subjects | 0 | 2

5. Secondary Outcome: Clinical Global Impression Scale of Improvement (CGI-I) Score at End of Double Blind Phase Relative to End of Open Label Phase (Baseline).
Description: The scale provides a global rating of illness improvement during the trial. The subject is rated relative to the clinician's past experience with other subjects who have the same diagnosis. The CGI-I scale is 1 question, and rates improvement compared with a baseline visit using a 7-point scale. The range of responses are from 1 (very much improved) through 7 (very much worse).
  A lower value is a better the outcome.
Time Frame: 2 weeks: End of open label phase (Baseline) at study day 84 to end of double blind treatment at study day 98.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aptensio XR | Placebo Comparator
Number analyzed (Participants) | 39 | 50
Participants
  1 = Very much improved | 6 | 5
  2 = Much improved | 8 | 6
  3 = Minimally improved | 3 | 4
  4 = No change | 11 | 13
  5 = Minimally worse | 4 | 1
  6 = Much worse | 6 | 16
  7 = Very much worse | 1 | 5

6. Secondary Outcome: Conners Early Childhood Behavior - Parent (Short) (EC BEH-P(S)) Change in T-score From End of Open Label Phase (Baseline) to End of Double Blind
Description: Conners EC BEH-P(S) is an assessment tool used to obtain a parent's observations about his/her child's behavior. This tool is designed to assess a range of behavioral, emotional, & social issues in young children. The tool consists of 47 items, responses to which are summarized in 6 behavioral scales & 2 validity scales.
  Items on Conners assessment are rated on a Likert scale ranging from 0-3. The ratings were converted to raw item scores. Raw item scores were grouped, standardized, and/or compared to lookup tables for interpretation. Assessments were presented as T-scores: item raw scores for a given scale are added together; this raw sum is compared to age- and gender-matched normative data and converted to a T-score. Higher scores indicate higher concerns. T-score is a standard score with a mean of 50 and standard deviation of 10. Note that Conners assessments do not use T-scores greater than 90; raw scores that produce extremely high T-scores are reported as ''T-score >= 90."
Time Frame: 2 weeks: End of open label phase (Baseline) at study day 84 to end of double blind treatment at study day 98.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aptensio XR | Placebo Comparator
Number analyzed (Participants) | 39 | 50
T-score
  Inattention/Hyperactivity | 1.92 (11.412) | 7.73 (15.067)
  Defiant/Aggressive Behaviors | 1.00 (11.016) | 3.67 (11.033)
  Social Functioning / Atypical Behaviors | 3.79 (10.437) | 3.83 (11.960)
  Anxiety | 1.89 (10.211) | -0.02 (8.299)
  Mood and Affect | 2.63 (11.780) | 5.13 (12.335)
  Physical Symptoms | 1.92 (13.200) | -0.15 (11.130)

ADVERSE EVENTS:
Time Frame: The AE-reporting period for this trial began at the Screening visit and ended with the 2-week follow-up phone call at end of study, up to 20 weeks.
Description: AEs were summarized for any exposure to Aptensio XR during the open-label treatment phase, and for each treatment (i.e., Aptensio XR or placebo) in the double-blind phase.
Arm/Group | Open-label Treatment Phase | Aptensio XR | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/40 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/119 | 0/40 | 0/50
Other Adverse Events (participants affected / at risk) | 82/119 | 6/40 | 2/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Treatment Phase (N=119) | Aptensio XR (N=40) | Placebo Comparator (N=50)
Campylobacter infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Treatment Phase (N=119) | Aptensio XR (N=40) | Placebo Comparator (N=50)
Insomnia (Psychiatric disorders) | 18 | 0 | 0
Irritability (Psychiatric disorders) | 17 | 0 | 0
Emotional Disorder (Psychiatric disorders) | 14 | 0 | 1
Affect lability (Psychiatric disorders) | 12 | 0 | 0
Initial insomnia (Psychiatric disorders) | 8 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 25 | 1 | 0
Weight decreased (Investigations) | 21 | 0 | 0
Hypertension (Vascular disorders) | 16 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 8 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 0 | 1
Headache (Nervous system disorders) | 9 | 0 | 0
Pyrexia (General disorders) | 7 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT02683265/Prot_SAP_000.pdf